CLINICAL TRIAL: NCT06420895
Title: Setting up a Health Data Warehouse on Aortic Insufficiency
Brief Title: Health Data Warehouse on Aortic Insufficiency
Acronym: EDS-AI
Status: Active, not recruiting | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: EDS-2023-02
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Aortic Insufficiency; Heart Valve Diseases
Keywords: aortic insufficiency; valvulopathy; Transthoracic echocardiogram; ultrasound; transesophageal echocardiogram; Data Warehouse
MeSH Terms: conditions — Aortic Valve Insufficiency; Heart Valve Diseases | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group of patients with aortic insufficiency: Patients already assessed at GHICL's Valvulopathy Centre from 2011 to October 2023 will be identified retrospectively, by queries based on keywords and/or diagnostic codes in echocardiography interpretation software (Viewpoint/EchoPAC, ISCV). GHICL's Medical Information Department will also be involved.
  Interventions: Other: Clinical follow-up; Other: Transthoracic Echocardiogram (TTE); Other: Magnetic resonance imaging (MRI); Other: Transesophageal echocardiogram (TEE)

INTERVENTIONS:
Other: Clinical follow-up — Clinical follow-up of patients
Other: Transthoracic Echocardiogram (TTE) — Transthoracic Echocardiogram
Other: Magnetic resonance imaging (MRI) — Magnetic resonance imaging
Other: Transesophageal echocardiogram (TEE) — Transesophageal echocardiogram

SUMMARY:
This project aims to create a data warehouse based on care data of patients with an aortic insufficiency admitted to the Groupement des Hôpitaux de l'Institut Catholique de Lille (GHICL) since 2011.

The aim is to enable the utilisation of this data for research purposes.

DETAILED DESCRIPTION:
All eligible patients will be informed about the collection of their data during their care at the Valvulopathies Center of Groupement des Hopitaux de l'Institut Catholique de Lille (GHICL). Their consent will be needed for the inclusion.

Data will be collected exclusively by the person responsible for implementing the data processing and his/her authorised staff. For all patients, data will be collected retrospectively, based on medical records (electronic or paper), and information available on the various care software linked to the patient's file. There will not be changes in the the patient's care.

At the GHICL Valvulopathy Centre, in accordance with European recommendations, patients with aortic insufficiency are monitored as follows, depending on the severity of the pathology:

* Minimal aortic insufficiency: follow-up every 3-5 years (approximately) including clinical examination and transthoracic echocardiogram (TTE)
* Moderate/medium aortic insufficiency: follow-up every 1-2 years with clinical examination, laboratory tests and TTE.
* Significant aortic insufficiency: follow-up every 6-12 months including a clinical examination, a biological assessment and a c+/- TTE coupled with an exercise test.
* Cardiac Magnetic Resonance Imaging (MRI) indicated as a second-line procedure after TTE in cases of moderate/medium aortic insufficiency with arguments or doubts about an underestimation of the severity of the aortic insufficiency on TTE, aortic insufficiency of undetermined quantification on TTE, or significant aortic insufficiency on TTE to confirm the severity using a multiparametric approach.
* TEE (transesophageal echocardiogram) is indicated as 2nd line after TTE in cases of significant aortic insufficiency as part of the preoperative work-up or moderate/undetermined aortic insufficiency on TTE.

The choice between cardiac MRI or TEE, or both, as second-line treatment after TEE, is left to the clinician in current practice, in accordance with the recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >= 18 years)
* Cared for at GHICL Since 1st January 2011
* With chronic aortic insufficiency of any grade.

Exclusion Criteria:

* Patients who have undergone prosthetic aortic valve surgery prior to diagnostic transthoracic echocardiography
* Patients with acute heart failure
* Patients with an intracardiac shunt or other complex congenital heart disease or obstructive hypertrophic cardiomyopathy
* Patients with aortic prosthesis
* Patients with active endocarditis or sequelae < 6 months old
* Patients under legal protection
* Patient who refused to take part in the study
* Patients with other than minimal left heart valve disease (with the exception of secondary mitral insufficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already assessed at GHICL's Valvulopathy Centre from 2011 to October 2023 will be identified retrospectively, by queries based on keywords and/or diagnostic codes in echocardiography interpretation software (Viewpoint/EchoPAC, ISCV). GHICL's Medical Information Department (DIM) will also be involved.
  Eligible patients assessed at GHICL's Valvulopathy Centre after the implementation of the repository (from November 2023) will be identified by the cardiologist as and when required.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with aortic insufficiency | one day
  Whereas this is a data mining process, no description can be provided

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Altes, MD, Principal Investigator — altes.alexandre@ghicl.net

IPD SHARING:
Plan to Share IPD: Undecided